CLINICAL TRIAL: NCT06832748
Title: Feasibility of a Virtual Reality Based Sensorimotor Training Intervention for Patients with Chronic Traumatic Neck Pain
Brief Title: Neck Movement Training in a Virtual Reality Headset for People with Neck Pain - a Feasibility Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luleå Tekniska Universitet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPM Dnr 2024-07490-01; CIV 24-08-048898 (Other: Swedish medical products agency)
Record Dates: First submitted 2025-01-31; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Neck Pain
Keywords: neck pain; virtual reality; VR; sensorimotor training; pilot RCT; endurance training; whiplash injuries; feasibility studies; randomized controlled trial
MeSH Terms: conditions — Neck Pain; Whiplash Injuries

STUDY DESIGN:
Intervention Model Description: This is a feasibility study and pilot randomized controlled trial (RCT). The study will gain knowledge of feasibility of the intervention before a future full scale RCT. The study has a quantitative part to assess the feasibility of the VR-intervention, and to obtain initial measures of possible intervention effects for future sample size calculation when compared to a more traditional rehab intervention. It has also a qualitative part including interviews with the participants in the VR-group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR neck training group (10 participants) (Experimental): 10 participants will use a VR headsets and perform training targeting the neck sensorimotor function. The patient interacts through head movements, and perform tasks in the VR environment.
  Interventions: Other: VR neck training
- Endurance neck training group (10 participants) (Active Comparator): 10 participants will perform endurance training for the neck and shoulder region, with body weight, rubber bands, and free weights.
  Interventions: Other: Endurance neck training

INTERVENTIONS:
Other: VR neck training — VR intervention 8 weeks. A VR headset is used for assessment and training of sensorimotor functions of the neck. The VR headset has a built-in sensor which can measure movements and give objective test and training results. The results serve as a guide for tailored home-based training programs, also performed with the VR headset in the experimental group. The participant performs the training at home, 15-20 minutes/day 5 days/week, initiallay divided into 3 sessions of 5 minutes each, while progression may lead to longer but fewer sessions. The program is individually tailored to target specific sensorimotor disturbances, and progressed during the intervention to increase the challenge. Participants will have video consultations with their physiotherapist once a week for the first 4 weeks, and every second week for the final 4 weeks. This can be adjusted to fit the participants needs. The VR is a novel technology, and this particular VR based training is not yet evaluated in research.
  Arms: VR neck training group (10 participants)
Other: Endurance neck training — An 8-week traditional endurance neck training intervention. The training program consists of neck and shoulder exercises performed with body weight, rubber bands, and free weights. The training is carried out at home, 15-20 minutes per day, 5 days a week. The training is individualized and progressed during the intervention. Participants will have video consultations with their physiotherapist once a week for the first 4 weeks, and then every second week for the final 4 weeks. This can be adjusted to fit the participants needs. This intervention is often used in the clinic and has been evaluated in several research studies with good results to reduce neck pain. However, its effects on sensorimotor functions have been less evaluated. Also, its effects compared to novel VR-training still needs to be evaluated.
  Arms: Endurance neck training group (10 participants)

SUMMARY:
The goal of this clinical trial is to learn if a virtual reality (VR) intervention for people with chronic neck pain is feasible. The main questions it aims to answer are:

Is it possible to perform a future full-scale randomized controlled trial (RCT) with a remotely supervised VR-based intervention for people with chronic neck pain?

How do people with neck pain experience using VR in a home-based training intervention?

Researchers will investigate if aspects of a full-scale RCT is feasible. This includes how well the recruitment of participants worked, retention during the intervention, compliance to training program, adverse events, and experience using the VR during training. The study will also investigate initial indication of benefit of the VR intervention, such as effects on pain and function.

Participants will be randomly assigned to either a VR neck training group or an endurance training group. Both groups will perform a training program for 8 weeks with weekly follow ups with their physiotherapist via online meetings.

DETAILED DESCRIPTION:
Title: Feasibility of a Virtual Reality-Based Sensorimotor Training Intervention for Patients with Chronic Traumatic Neck Pain

Background: Neck pain is very common, leading to reduced function and quality of life, and is costly for healthcare and society due to sick leave and productivity loss. The cause of neck pain is often unclear, with no visible structural damage. Persistent neck pain (lasting more than 3 months) and recurrent episodes are complex and not fully understood. Research suggests impaired sensorimotor control as a contributing factor.

Sensorimotor control involves neck movement control, awareness of head position, quick reaction to stimuli, and good neck mobility. These functions are crucial for daily activities (e.g., moving our body, riding a bike, driving a car), and maintaining body stability. Research has shown that these functions often are impaired in people with neck pain. Training these functions can reduce pain and improve function.

Virtual Reality (VR) technology, especially VR headsets, allows objective assessment of neck sensorimotor functions, crucial for personalized training to reduce pain and improve function. VR can measure movement velocity and reaction time, previously only possible with advanced lab equipment. VR can be used in clinics and at home, showing high accuracy in assessing neck functions. It may also make training enjoyable, potentially improving adherence.

Aim: This study aims to assess the feasibility of a future large-scale randomized controlled trial (RCT) using a VR-based training program for chronic neck pain patients. It will explore various feasibility aspects to plan a well-conducted RCT and examine participants' experiences with VR. Aspects include participant recruitment, adherence to intervention, study protocol feasibility, experience of VR based intervention, and initial effects on pain and function. Data will also help calculate the required sample size for a future RCT.

Method: The study is a pilot RCT with 20 participants randomized into two groups: VR training or endurance training. A stratified randomization to get equal number of women/men in each group will be performed through a randomization program. Both groups will train at home for 8 weeks with digital follow-ups from a physiotherapist.

There will be 2 qualified physiotherapists, each treating 10 patients (5 in each group). The physiotherapists have solid clinical experience from primary health care. They have experience treating people with neck pain and prescribing sensorimotor exercises. The physiotherapists will conduct baseline and post-treatment measures of outcome variables. They will not be blinded to treatment allocation.

Patients and physiotherapists will not be blinded to treatments due to the interventions being self-revealing.

After the intervention, VR group participants will be interviewed about their VR experience.

Participants: The study will include individuals with chronic neck pain (lasting more than 3 months) caused or worsened by trauma (e.g., car accidents, falls).

Outcome: The study will result in two publications: one on quantitative feasibility data, and another on qualitative feasibility data (patient interviews).

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand verbal and written Swedish
* Persistent neck pain (>3 months)
* Neck pain onset (or acute worsening) in relation to trauma to the head or neck
* Neck disability index 20-60% or Numeric Rating Scale neck pain ≥ 3/10
* Impaired sensorimotor function of the neck (at least one of the sensorimotor tests must be impaired, i.e. below the norm values for the test in question). The following cut-off values are used:

Joint position sense test: > 4.5° absolute error in any of the four directions right rotation, left rotation, extension or flexion.

Movement sense test: >28 seconds to complete the zigzag pattern, or <2,5 norm value (i.e., accuracy in percentage divided by time in seconds).

Maximum velocity from the cervical reaction acuity test: < 100°/s. Range of motion in right rotation, left rotation, extension and flexion (added together): < 300°.

Exclusion Criteria:

* Cervical radiculopathy
* Neck surgery
* Fracture of the neck
* Neurological disease
* Vestibular disease
* Rheumatic disease
* Concussion where the person lost consciousness
* Uncorrected visual impairment
* Epilepsy
* Previous experience of severe symptoms (nausea/dizziness) when using VR headsets

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Recruitment time (weeks) | From enrollment to end of treatment (at 8 weeks)
  Time taken to recruit 20 participants. This will be measured in number of weeks.
Feasibility - Recruitment method | From enrollment to end of treatment (at 8 weeks)
  Which recruitment channels were effective to find participants? (physiotherapy clinics, social media channels, newspaper advertisement, other). This will be measured by asking the participants.
Feasibility - Adherence | Start of intervention to end of intervention at 8 weeks.
  Adherence rate to interventions. For the VR training group this is evaluated from the VR online portal training log. For the endurance training group this is evaluated from training diaries. This will be measured by number of completed training sessions and presented as percentage of prescribed dosage. A minimum of 70 % completed training sessions is considered acceptable.
  Adherence feasibility criteria: ≥ 70% Proceed, 60-69% Proceed with changes, <60% Do not proceed
Feasibility - Completion rate (drop out) | Start of intervention to end of intervention at 8 weeks.
  Number of participants completing the intervention. Intervention completion rate feasibility criteria: ≥ 85% proceed, 70-85% proceed with changes, <70% do not proceed.
Feasibility - Outcome measure completion rate | At 8 weeks
  Obtained outcome measures from participants completing the intervention. Outcome measure completion rate criteria: ≥ 85% Proceed, 70-85% Proceed with changes, <70% Do not proceed
Feasibility - Adverse events | From start of intervention to 8 weeks
  Number of adverse events and what character. Treating physiotherapists will record any adverse events during the intervention period.
Feasibility - Numeric Rating Scale (NRS) Simulator sickness intensity | Baseline and at end of intervention (at 8 weeks).
  Sickness intensity measured by the eleven-point Numeric Rating Scale (NRS), 0-10. The participants rate their sickness intensity right after completion of the test protocol, from no sickness (0) to worst imaginable sickness (10).
Feasibility - Participants experience using VR in neck training - Qualitative part | After completion of the 8 weeks VR-intervention, approximately within 2 weeks after completion.
  Participants experience using VR in the 8-week intervention. This information will be obtained from semi-structured interviews, e.g., questions about usability, digitally delivered intervention, video consultations with physiotherapists, information and support, pros and cons of intervention.

SECONDARY OUTCOMES:
Cervical joint position sense (JPS) test (performed in the VR headset) | Baseline and at end of intervention (at 8 weeks)
  Cervical JPS test assessed in the VR headset. The JPS test assesses the ability to sense the position of the neck and head (part of proprioception).
  With a dark VR screen (imitating being blindfolded), the task is to find neutral head position, perform a head movement, and reposition the head back to the neutral position as accurately as possible. The test is performed with 6 repetitions i right rotation, left rotation, extension and flexion respectively. The error from starting position to end position is measured in degrees. Absolute error is calculated as outcome measure.
Cervical reaction acuity (CRA) test - Reaction time milliseconds (performed in the VR headset) | Baseline and at end of intervention (at 8 weeks)
  CRA test assessed in the VR headset. A ball on the VR screen will move from the center to a random location. The task is to follow the ball as quickly as possible by moving the head to the center of the ball and staying in the center until a time circle counts down. The ball appears in the middle again, the participant moves their head back there and the next attempt begins. This will be repeated in random directions for 8 repetitions. Reaction time is measured in milliseconds, and defined as the time from the movement of the ball to the participant reaching 5% of their maximum velocity.
Cervical reaction acuity (CRA) test - Maximum velocity. (performed in the VR headset) | Baseline and at end of intervention (at 8 weeks)
  CRA test assessed in the VR headset. A ball on the VR screen will move from the center to a random location. The task is to follow the ball as quickly as possible by moving the head to the center of the ball and staying in the center until a time circle counts down. The ball appears in the middle again, the participant moves their head back there and the next attempt begins. This will be repeated in random directions for 8 repetitions. Maximum velocity per repetition is measured in degrees per seconds.
Cervical reaction acuity (CRA) test - Time to complete the task. (performed in the VR headset) | Baseline and at end of intervention (at 8 weeks)
  CRA test assessed in the VR headset. A ball on the VR screen will move from the center to a random location. The task is to follow the ball as quickly as possible by moving the head to the center of the ball and staying in the center until a time circle counts down. The ball appears in the middle again, the participant moves their head back there and the next attempt begins. This will be repeated in random directions for 8 repetitions. Time to complete the task is measured in seconds.
Cervical movement sense test (performed in the VR headset) | Baseline and at end of intervention (at 8 weeks)
  Cervical movement sense test assessed in the VR headset. With head movements, participant trace the lines of a zig zag pattern as accurately as possible to their self-chosen speed. Outcome measures are:
  * Accuracy in percentage representing the percentage of the time being on the line.
  * Time to complete the task.
  * Norm value (accuracy divided by time).
Cervical range of motion test (performed in the VR headset) | Baseline and at end of intervention (at 8 weeks)
  Maximum cervical range of motion in degrees is assessed in the VR headset for
  * right rotation
  * left rotation
  * extension
  * flexion
  * right lateral flexion
  * left lateral flexion
  * right diagonal extension
  * left diagonal extension
  * right diagonal flexion
  * left diagonal flexion
Postural sway in quiet stance (performed with the VR headset) | Baseline and at end of intervention (at 8 weeks)
  Postural sway assessed in the VR headset. Quiet stance with feet together and arms crossed over the chest. The task is to stand as still as possible for 30 seconds with eyes open and closed, respectively. Outcome measures are the total length of the sway path in cm and sway amplitude in cm in anterio-posterior and medio-lateral direction, respectively. Data will be normalized to the height of the person.
Cervical flexion endurance test | Baseline and at end of intervention (at 8 weeks)
  The participant lies in supine position, legs bent to 90 degrees. The chin is flexed while lifting the head and neck to about 2.5 cm above the surface. The test leader places one hand on the surface just below the participant's occiput to feel when the participant loses lift.
  The test ends if the participant touches the test leader's hand for more than one second or if the participant loses the flexion of the chin.
  Outcome measures are seconds.
Neck Disability Index (NDI) | Baseline and at end of intervention (at 8 weeks)
  A self-reported physical functioning questionnaire targeting pain intensity and how it interferes with daily activities. Maximum score is 50 where a higher score represents higher disability. The score is transformed to percentage, higher percentage representing higher disability.
Numeric Rating Scale (NRS) neck pain | Baseline and at end of intervention (at 8 weeks)
  Pain intensity measured by the eleven-point Numeric Rating Scale (NRS), 0-10. The participants rate their average pain intensity the previous 7 days, from no pain (0) to worst imaginable pain (10).
Numeric Rating Scale (NRS) dizziness | Baseline and at end of intervention (at 8 weeks)
  Dizziness intensity will be measured by the eleven-point Numeric Rating Scale (NRS), 0-10. The participants rate their average dizziness intensity the previous 7 days from 0=no dizziness to 10= worst imaginable dizziness.
Numeric Rating Scale (NRS) headache | Baseline and at end of intervention (at 8 weeks)
  Headache intensity will be measured by the eleven-point Numeric Rating Scale (NRS), 0-10. The participants rate their average headache intensity the previous 7 days from 0=no headache to 10=worst imaginable headache.
EQ-5D-5L | Baseline and at end of intervention (at 8 weeks)
  Euro Quality of life 5 Dimensions 5 Levels (EQ-5D-5L). This is a questionnaire measuring health related quality of life. It is made up of 5 questions concerning mobility, personal care, daily activities, pain and discomfort, and psychological function (anxiety/depression). Each question gives a score from 1-5 where 1 = no problem and 5 = major problems and gives a 5-digit score which relates to a health profile.
Tampa scale of kinesiophobia -short version 11 item (TSK-11) | Baseline and at end of intervention (at 8 weeks)
  Fear of movement questionnaire. It consists of 11 items, 1-4-point scale, where a higher score represents higher fear of movement.
Global perceived effect (GPE) | At end of intervention (at 8 weeks)
  The global perceived effect scale is used to measure how much the participants neck problem has changed since the start of the intervention. It is an 11-point scale where -5=Much worse 0=No change, and +5=Much better
Feasibility - Physiotherapists experience of the VR intervention- Measured with a questionnaire. | After all participants have completed post intervention assessments at the end of the intervention (at 8 weeks)
  Treating physiotherapists' experience of carrying out the VR intervention is evaluated with a questionnaire. It contains questions targeting aspects of the VR intervention, such as delivering the intervention remotely, advantages and disadvantages compared to traditional treatment with patient visits at a clinic, and usability aspects. The questionnaire comprises of nine 9-point Likert-scale questions, where 1 represents "strongly disagree" and 9 represents "strongly agree". Higher number indicate a more positive rating. Two open questions are included for comments about pros and cons of the VR-technology.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Röijezon, Professor, Study Chair — Luleå University of Technology. Department of Health, Education and Technology

IPD SHARING:
Plan to Share IPD: No
Due to sensitive data (health data) being collected.

REFERENCES:
- [Background] GBD 2016 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 328 diseases and injuries for 195 countries, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1211-1259. doi: 10.1016/S0140-6736(17)32154-2. PMID 28919117
- [Background] Treleaven J. Sensorimotor disturbances in neck disorders affecting postural stability, head and eye movement control. Man Ther. 2008 Feb;13(1):2-11. doi: 10.1016/j.math.2007.06.003. Epub 2007 Aug 16. PMID 17702636
- [Background] Safiri S, Kolahi AA, Hoy D, Buchbinder R, Mansournia MA, Bettampadi D, Ashrafi-Asgarabad A, Almasi-Hashiani A, Smith E, Sepidarkish M, Cross M, Qorbani M, Moradi-Lakeh M, Woolf AD, March L, Collins G, Ferreira ML. Global, regional, and national burden of neck pain in the general population, 1990-2017: systematic analysis of the Global Burden of Disease Study 2017. BMJ. 2020 Mar 26;368:m791. doi: 10.1136/bmj.m791. PMID 32217608
- [Background] Sjolander P, Michaelson P, Jaric S, Djupsjobacka M. Sensorimotor disturbances in chronic neck pain--range of motion, peak velocity, smoothness of movement, and repositioning acuity. Man Ther. 2008 May;13(2):122-31. doi: 10.1016/j.math.2006.10.002. Epub 2007 Jan 2. PMID 17197230
- [Background] Sarig Bahat H, Croft K, Carter C, Hoddinott A, Sprecher E, Treleaven J. Remote kinematic training for patients with chronic neck pain: a randomised controlled trial. Eur Spine J. 2018 Jun;27(6):1309-1323. doi: 10.1007/s00586-017-5323-0. Epub 2017 Oct 10. PMID 29018956
- [Background] Sarig Bahat H, Chen X, Reznik D, Kodesh E, Treleaven J. Interactive cervical motion kinematics: sensitivity, specificity and clinically significant values for identifying kinematic impairments in patients with chronic neck pain. Man Ther. 2015 Apr;20(2):295-302. doi: 10.1016/j.math.2014.10.002. Epub 2014 Oct 14. PMID 25456272
- [Background] Roijezon U, Djupsjobacka M, Bjorklund M, Hager-Ross C, Grip H, Liebermann DG. Kinematics of fast cervical rotations in persons with chronic neck pain: a cross-sectional and reliability study. BMC Musculoskelet Disord. 2010 Sep 27;11:222. doi: 10.1186/1471-2474-11-222. PMID 20875135
- [Background] Roijezon U, Clark NC, Treleaven J. Proprioception in musculoskeletal rehabilitation. Part 1: Basic science and principles of assessment and clinical interventions. Man Ther. 2015 Jun;20(3):368-77. doi: 10.1016/j.math.2015.01.008. Epub 2015 Jan 29. PMID 25703454
- [Background] Qu N, Tian H, De Martino E, Zhang B. Neck Pain: Do We Know Enough About the Sensorimotor Control System? Front Comput Neurosci. 2022 Jul 15;16:946514. doi: 10.3389/fncom.2022.946514. eCollection 2022. PMID 35910451
- [Background] Peng B, Yang L, Li Y, Liu T, Liu Y. Cervical Proprioception Impairment in Neck Pain-Pathophysiology, Clinical Evaluation, and Management: A Narrative Review. Pain Ther. 2021 Jun;10(1):143-164. doi: 10.1007/s40122-020-00230-z. Epub 2021 Jan 12. PMID 33464539
- [Background] Jull G, Falla D, Treleaven J, Hodges P, Vicenzino B. Retraining cervical joint position sense: the effect of two exercise regimes. J Orthop Res. 2007 Mar;25(3):404-12. doi: 10.1002/jor.20220. PMID 17143898
- [Background] Moghaddas D, de Zoete RMJ, Edwards S, Snodgrass SJ. Differences in the kinematics of the cervical and thoracic spine during functional movement in individuals with or without chronic neck pain: a systematic review. Physiotherapy. 2019 Dec;105(4):421-433. doi: 10.1016/j.physio.2019.01.007. Epub 2019 Jan 21. PMID 31005251
- [Background] Malfliet A, Kregel J, Cagnie B, Kuipers M, Dolphens M, Roussel N, Meeus M, Danneels L, Bramer WM, Nijs J. Lack of evidence for central sensitization in idiopathic, non-traumatic neck pain: a systematic review. Pain Physician. 2015 May-Jun;18(3):223-36. PMID 26000666
- [Background] Kristjansson E, Treleaven J. Sensorimotor function and dizziness in neck pain: implications for assessment and management. J Orthop Sports Phys Ther. 2009 May;39(5):364-77. doi: 10.2519/jospt.2009.2834. PMID 19411769
- [Background] Kristjansson E, Bjornsdottir SV, Oddsdottir GL. The long-term course of deficient cervical kinaesthesia following a whiplash injury has a tendency to seek a physiological homeostasis. A prospective study. Man Ther. 2016 Apr;22:196-201. doi: 10.1016/j.math.2015.12.008. Epub 2015 Dec 23. PMID 26778601
- [Background] Ernst MJ, Williams L, Werner IM, Crawford RJ, Treleaven J. Clinical assessment of cervical movement sense in those with neck pain compared to asymptomatic individuals. Musculoskelet Sci Pract. 2019 Oct;43:64-69. doi: 10.1016/j.msksp.2019.06.006. Epub 2019 Jul 2. PMID 31277033
- [Background] Dieleman JL, Cao J, Chapin A, Chen C, Li Z, Liu A, Horst C, Kaldjian A, Matyasz T, Scott KW, Bui AL, Campbell M, Duber HC, Dunn AC, Flaxman AD, Fitzmaurice C, Naghavi M, Sadat N, Shieh P, Squires E, Yeung K, Murray CJL. US Health Care Spending by Payer and Health Condition, 1996-2016. JAMA. 2020 Mar 3;323(9):863-884. doi: 10.1001/jama.2020.0734. PMID 32125402
- [Background] Della Casa E, Affolter Helbling J, Meichtry A, Luomajoki H, Kool J. Head-eye movement control tests in patients with chronic neck pain; inter-observer reliability and discriminative validity. BMC Musculoskelet Disord. 2014 Jan 14;15:16. doi: 10.1186/1471-2474-15-16. PMID 24423109
- [Background] de Vries J, Ischebeck BK, Voogt LP, van der Geest JN, Janssen M, Frens MA, Kleinrensink GJ. Joint position sense error in people with neck pain: A systematic review. Man Ther. 2015 Dec;20(6):736-44. doi: 10.1016/j.math.2015.04.015. Epub 2015 May 2. PMID 25983238
- [Background] De Pauw R, Van Looveren E, Lenoir D, Danneels L, Cagnie B. Reliability and discriminative validity of a screening tool for the assessment of neuromuscular control and movement control in patients with neck pain and healthy individuals. Disabil Rehabil. 2022 Jan;44(1):139-147. doi: 10.1080/09638288.2020.1760948. Epub 2020 Jun 1. PMID 32478587
- [Background] Blanpied PR, Gross AR, Elliott JM, Devaney LL, Clewley D, Walton DM, Sparks C, Robertson EK. Neck Pain: Revision 2017. J Orthop Sports Phys Ther. 2017 Jul;47(7):A1-A83. doi: 10.2519/jospt.2017.0302. PMID 28666405